CLINICAL TRIAL: NCT04113434
Title: Linking Endotypes and Outcomes in Pediatric Acute Respiratory Distress Syndrome
Acronym: LEOPARDS
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Akron Children's Hospital (Other); Children's Hospital and Health System Foundation, Wisconsin (Other); Children's Hospital Medical Center, Cincinnati (Other); Children's Mercy Hospital Kansas City (Other); Milton S. Hershey Medical Center (Other); Nationwide Children's Hospital (Other); Nicklaus Children's Hospital (Unknown); Indiana University (Other); Cooperman Barnabas Medical Center (Unknown); Baylor College of Medicine (Other); Columbia University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Arkansas Children's Hospital Research Institute (Other); Children's Healthcare of Atlanta (Other); Children's Hospital Colorado (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 19-016271; R01HL148054 (NIH)
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress Syndrome; ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall goal of the study is to risk stratify pediatric Acute Respiratory Distress Syndrome (ARDS) patients and to identify sub-phenotypes with shared biology in order to appropriately target therapies in future trials. This is a prospective, multicenter study of 500 intubated children with ARDS, with planned blood collection within 24 hours of ARDS onset and subsequent measurement of plasma protein biomarkers and peripheral blood gene expression.

DETAILED DESCRIPTION:
Investigators will measure pre-determined biomarkers with known or suspected association with ARDS severity or outcome. Simultaneously, investigators will measure gene expression of peripheral blood. Both plasma biomarkers and gene expression profiles will be analyzed using various machine learning techniques, including classification and regression tree, latent class analysis, and hierarchical clustering with the goal of identifying sub-phenotypes of ARDS. These sub-phenotypes will be examined for association with outcome (primary is 28-day mortality), and explicitly tested for variation in response to exogenous treatments (e.g., corticosteroids).

ELIGIBILITY:
Inclusion Criteria:

1. acute (≤ 7 days of risk factor) respiratory failure requiring invasive mechanical ventilation
2. age > 44 weeks corrected gestational age and < 17.5 years
3. invasive mechanical ventilation via endotracheal tube
4. bilateral infiltrates on chest radiograph
5. oxygenation index (OI) ≥ 4; or oxygen saturation index (OSI) ≥ 5 on 2 consecutive measurements at least 4 hours apart but < 24 hours apart
6. invasively ventilated ≤ 7 days before meeting above radiographic and oxygenation criteria

Exclusion Criteria:

1. weight < 3 kilograms
2. cyanotic congenital heart disease (other than Patent Foramen Ovale (PFO) or Patent Ductus Arteriosus (PDA))
3. tracheostomy at time of screening
4. invasively ventilated for > 7 days when meet ARDS criteria above
5. cardiac failure as predominant cause of respiratory failure
6. primary obstructive airway disease (asthma, bronchiolitis) by judgement of clinician as the primary cause of respiratory failure
7. alternative known chronic lung disease as cause of respiratory failure (cystic fibrosis, eosinophilic pneumonia, interstitial pneumonitis, pulmonary hemosiderosis, cryptogenic organizing pneumonia)
8. severe neurologic morbidity not expected to survive > 72 hours
9. any limitations of care at time of screening
10. previous enrollment in this study

Ages: 44 Weeks to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants to adolescents between the ages of 44 weeks and 17.5 years, who are admitted to PICU for acute respiratory failure requiring invasive mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
28 Day Mortality in Pediatric ARDS. | 28 days
  28 day all cause mortality.
Presence of two or more endotypes in Pediatric ARDS. | Within 24 hours of ARDS onset
  Stratify pediatric ARDS into sub-phenotypes using a known 100-gene expression-based classifier to group subjects according to shared underlying biology.
Occurrence of de novo sub-phenotypes in pediatric ARDS using biomarkers and whole genome transcriptomics of peripheral blood. | Within 24 hours of ARDS onset.
  Occurrence of de novo sub-phenotypes in pediatric ARDS using 12 protein biomarkers and whole genome transcriptomics of peripheral blood.

SECONDARY OUTCOMES:
ventilator-free days at 28 days. | 28 days
  composite endpoint of days alive and free of mechanical ventilation by day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Nadir Yehya, M.D., Principal Investigator — Children's Hospital of Philadelphia
Locations (16):
- United States (16):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Colorado, Aurora, Colorado
  - Variety Children's Hospital D/B/A Nicklaus Children's Hospital, Miami, Florida
  - Children's Healthcare of Atlanta - Emory, Atlanta, Georgia
  - Riley Children's at Indiana University Health, Indianapolis, Indiana
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Cooperman Barnabas Medical Center, Livingston, New Jersey
  - Columbia University Medical Center, New York, New York
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital / Baylor College of Medicine, Houston, Texas
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Specific consent will be obtained to store blood and use data for future research. We will share data with the research community using the Biologic Specimen and Data Repository Information Coordinating Center (BioLINCC) program at NHLBI, and we will follow suggested guidelines for de-identifying the data (coding of site IDs, conversion of dates to study days).
  Pursuant to the NIH policy, all data obtained from this proposal will be made available for research by qualified individuals within the scientific community after publication of the proposed studies. Gene expression data from Aims 2 and 3 will be made available simultaneous with publication of the results of these aims by uploading to the Gene Expression Omnibus. For dissemination of plasma biomarker results and the associated clinical dataset, we will use BioLINCC program at NHLBI, with release of a de-identified dataset with untraceable identifiers within 2 years of publication of the main manuscript.
Supporting Information: Study Protocol, ICF
Time Frame: Gene expression data will be released to Gene Expression Omnibus simultaneously with the publication of the data. Biomarker data will be released within 2 years of publication of the main manuscript.
Access Criteria: We will follow NHLBI's guidelines for accessing BioLINCC data.

REFERENCES:
- [Derived] Whitney JE, Johnson GM, Varisco BM, Raby BA, Yehya N. Biomarker-Based Risk Stratification Tool in Pediatric Acute Respiratory Distress Syndrome: Single-Center, Longitudinal Validation in a 2014-2019 Cohort. Pediatr Crit Care Med. 2024 Jul 1;25(7):599-608. doi: 10.1097/PCC.0000000000003512. Epub 2024 Apr 9. PMID 38591949